CLINICAL TRIAL: NCT05935761
Title: Investigating Novel Interventions for Low Back Pain in US Military Veterans: A Randomized Controlled Adaptive Phase II Trial
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NURP-004-22F; I01CX002667-01 (NIH)
Record Dates: First submitted 2023-06-28; First posted 2023-07-07 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Chronic Low Back Pain
Keywords: neurosteroid; pregnenolone; DHEA; Veteran; Pain; Back
MeSH Terms: conditions — Pain | interventions — Pregnenolone; Dehydroepiandrosterone

STUDY DESIGN:
Intervention Model Description: Randomized, double-blind, placebo controlled trial.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-blinded study, all are blinded except for the research pharmacist who creates the randomization schedule.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Pregnenolone (Active Comparator): Pregnenolone dosing will begin at 500mg/day x 7 days, and will increase by 500mg each following week as tolerated (to a potential maximum dose 2000mg/day).
  Interventions: Drug: Pregnenolone
- DHEA (Active Comparator): DHEA dosing will begin at 100mg/day x 7 days, and will increase by 100mg each following week as tolerated (to a potential maximum dose 400mg/day).
  Interventions: Drug: DHEA
- Placebo (Placebo Comparator): Same as active comparator arms, except placebo dispensed
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Pregnenolone — Pregnenolone dosing will begin at 500mg/day x 7 days, and will increase by 500mg each following week as tolerated (to a potential maximum dose 2000mg/day).
  Arms: Pregnenolone
Drug: DHEA — DHEA dosing will begin at 100mg/day x 7 days, and will increase by 100mg each following week as tolerated (to a potential maximum dose 400mg/day).
  Arms: DHEA
Drug: Placebo — Same as active comparator arms, except placebo dispensed
  Arms: Placebo

SUMMARY:
Chronic pain symptoms are very common among U.S. Military Veterans and have a profound negative impact on mental health symptoms and quality of life, in addition to increasing risk for suicidal ideation and suicidal behaviors. There are currently extremely few safe and effective pharmacological treatments for chronic pain disorders, and the clinical need to develop new therapeutics for pain has never been more urgent. Fueled by the worsening opioid crisis and further exacerbated by the COVID-19 pandemic, opioid and other drug overdose deaths have climbed to staggeringly high levels. The rapid development of medications for the management of chronic pain conditions that are safe, well-tolerated, efficacious and non-addicting is thus of paramount importance. The two neurosteroid candidates to be investigated in this trial are naturally occurring molecules enriched in human brain and potentially ideal candidates for safe and effective chronic pain treatment.

DETAILED DESCRIPTION:
Pain is one of the most common reasons that Americans seek medical care, with more than 50 million Americans reporting pain that is chronic (CDC NHIS data) and almost 20 million Americans reporting high impact pain that affects major life activities (Nahin, 2015). Chronic pain conditions disproportionately impact U.S. Military Veterans, and back pain is one of the most common diagnoses among Iraq/Afghanistan-era Veterans. The often-debilitating sequelae of chronic low back pain profoundly impacts quality of life and function in a very large number of Veterans and is substantial risk factor for the development or worsening of depression, anxiety and suicidal ideation. Commonly used treatments for pain include long-term opioid use, which is frequently suboptimal and has played a substantial role in the recent surge of opioid-related addiction and deaths. Non-opioid pharmacological interventions that maximize analgesia and minimize adverse outcomes are thus of critical national importance.

Neurosteroids exhibit pleiotropic actions that are highly relevant to central nervous system conditions, including pain disorders. Both preclinical and clinical studies provide strong evidence for the role of neurosteroids in pain. Among other similar studies, the investigators' laboratory has also demonstrated that allopregnanolone levels are reduced in Veterans reporting low back pain and chest pain. Moreover, the recently completed randomized clinical trial (RCT) demonstrated that Veterans randomized to pregnenolone (an endogenous precursor of allopregnanolone) demonstrated significant reduction in low back pain compared to placebo (Naylor et al 2020). The highest dose of pregnenolone resulted in the greatest improvements in pain intensity ratings but the investigators' data suggested that higher doses of this molecule may be even more efficacious. Thus, an RCT to optimize dosing of pregnenolone is warranted. Furthermore, dehydroepiandrosterone (DHEA) is another neurosteroid that has been implicated in pain. The investigators' laboratory (and others) demonstrates that DHEA levels are generally inversely associated with pain and the preliminary data indicate that supplementation with DHEA is associated with a reduction in pain symptoms. Administration of DHEA could thus also represent a novel therapeutic intervention for chronic pain symptoms. The investigators therefore propose to utilize an efficient and informative adaptive trial design to evaluate the efficacy and safety of these two promising molecules for the treatment of chronic low back pain.

Specific Aim 1: To conduct a Phase II adaptive randomized, double-blind, placebo-controlled trial with flexible dosing of pregnenolone, DHEA or placebo (1:1:1 randomization) to highest well-tolerated doses in 108 Veterans with chronic low back pain who served in the U.S. Military. Safety and efficacy will be determined for each chronic low back pain intervention over the course of 4 weeks (total study duration is 6 weeks). Hypothesis 1: Based on the investigators' previously published RCT showing that 500 mg of pregnenolone significantly reduces low back pain, it's hypothesize the investigators will replicate these positive findings with the pregnenolone 500 mg dosing strategy and that pregnenolone at higher doses of 1,000 mg and 2,000 mg per day will result in even greater improvements in low back pain Hypothesis 2: DHEA levels at baseline and post-treatment will predict therapeutic response and higher doses will result in greater improvement in low back pain. Hypothesis 3: Pregnenolone and DHEA will be safe and well-tolerated in this adaptive clinical trial design using flexible dosing.

Specific Aim 2: To conduct biomarker candidate investigations quantifying pregnenolone, DHEA and their neurosteroid metabolite levels (allopregnanolone, others) in serum at baseline, during treatment and post-treatment with pregnenolone and DHEA using highly sensitive and specific mass spectrometry-based methodologies (GC/MS/MS) in order to: a.) characterize the metabolic profile and pharmacokinetics of pregnenolone and DHEA and b.) identify predictors of therapeutic response (potentially yielding valuable dosing information and identifying windows of optimal therapeutic efficacy). Hypothesis: Based on the preliminary candidate biomarker data, the investigators hypothesize that changes in pregnenolone, pregnenolone metabolites, DHEA and DHEA metabolite levels post-treatment will be predictive of therapeutic response and identify optimal therapeutic ranges.

As chronic low back pain conditions significantly impact Veterans, there is an urgent need for the development of pharmacological treatments that are safe, efficacious and non-habit forming. The proposed adaptive platform RCT would thus provide pivotal evidence to optimize treatment in pain disorders for Veterans that could be easily translated to active duty and civilian populations. This RCT thus potentially represents a therapeutic breakthrough for the treatment of pain and may also have the added benefit of mitigating other commonly co-occurring symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Veterans, 18-65 years of age with chronic low back pain.
* Based on medical history and medical records, have low back pain (Thoracic Vertebrae 6 or below) present on most days for the preceding 6 months or longer, and fulfill all disease diagnostic criteria (please see disease diagnostic criteria below).
* Have a weekly mean of 24-hour average pain score 4 at baseline.
* Negative pregnancy test if female. Sexually active subjects are required to use a medically acceptable form of birth control if they are of childbearing potential and could become pregnant during the study. A medically acceptable form of birth control includes non-hormonal intrauterine devices, surgical sterilization, or double barrier methods (e.g. diaphragm with contraceptive jelly, condom with contraceptive foam, cervical caps with contraceptive jelly). Sexual abstinence with agreement to continue abstinence or to use a medically acceptable method of contraception (as listed above) should sexual activity occur is permissible.
* No change in medications less than 4 weeks before baseline.
* No anticipated need to alter psychotropic or pain medications for the 6-wk study duration (as determined by study physician's review of records and/or discussion with prescribing physician).
* Ability to fully participate in the informed consent process.

Exclusion Criteria:

* Unstable medical or neurological illness, including seizures, renal impairment or cerebral vascular accident (CVA).
* Use of oral contraceptives or other hormonal supplements-this is out of caution, as it is unknown if the study medications would impact the efficacy of hormonal contraception.
* Significant suicidal or homicidal ideation that necessitates intervention.
* Daily use of long or short-acting narcotic medications (PRN use will be considered).
* Current DSM-5 diagnosis of bipolar disorder, schizophrenia, or other psychotic disorder, or cognitive disorder due to a general medical condition.
* Female participants who are pregnant or breast-feeding.
* Known allergy to study medication.
* History of moderate or severe TBI (mild TBI is permissible).
* DSM-5 criteria met for alcohol and/or other substance abuse or dependence within past three months (excludes caffeine and nicotine).
* Have received epidural steroids, facet block, nerve block or other invasive procedures aimed to reduce low back pain within the past 3 months prior to Visit 1.
* Have ongoing or anticipated disability compensation or litigation issues, in the best judgment of the investigator.
* Have a presence of any factors/conditions, medical or other, that in the judgment of the investigator may interfere with performance of study outcome measures, such as treatment-refractory history.
* Have serious or unstable cardiovascular, hepatic, renal, metabolic, respiratory, or hematologic illness, symptomatic peripheral vascular disease, or other medical condition or psychiatric conditions that, in the opinion of investigator and study physician, would compromise participation or be likely to lead to hospitalization during the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2029-10-01 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Pain Numerical Rating Scale (0-10) Change | Visit 1 (Week 1/screening), Visit 2 (Week 2/Randomization/Baseline), Visit 3 (Week 3), Visit 4 (Week 4), Visit 5 (Week 5), Visit 6 (Week 6)
  Weekly mean of the 24-hour average pain severity scores recorded daily on an 11-point numerical rating scale, an ordinal scale ranging from 0 (no pain) to 10 (worst possible pain).

SECONDARY OUTCOMES:
Brief Pain Inventory | Visit 1 (Week 1/screening), Visit 2 (Week 2/Randomization/Baseline), Visit 3 (Week 3), Visit 4 (Week 4), Visit 5 (Week 5), Visit 6 (Week 6)
  The BPI is a self-reported scale that measures the severity of pain and the interference of pain on function. The scores range from 0 (no pain) to 10 (pain as severe as you can imagine). There are 4 questions assessing worst pain, least pain, average pain in the past 24 hours, and the pain right now. The Interference scores range from 0 (does not interfere) to 10 (completely interferes). There are 7 questions assessing the interference of pain in the past 24 hours for general activity, mood, walking ability, normal work, relations with other people, sleep, and enjoyment of life. Questions from the BPI will be asked at each study visit.

OTHER OUTCOMES:
Beck Depression Inventory, 2nd Edition | Visit 1 (Week 1/screening), Visit 2 (Week 2/Randomization/Baseline), Visit 3 (Week 3), Visit 4 (Week 4), Visit 5 (Week 5), Visit 6 (Week 6)
  The BDI-II is a 21-item self-reported questionnaire which measures the existence and severity of symptoms of depression. Each of the 21 items on BDI-II tool represents a depressive symptom. The symptoms are each scored on a 4-point Likert scale of 0 to 3 (0=symptom is absent; 3=symptom is severe). Scores for each symptom are added up to obtain the total scores for all 21 items. Total score ranges from 0-63; of which 0-8 is considered no depression, 0-13 is minimal depression, 14-19 is mild depression, 20-28 is moderate depression and 29-63 is severe depression.
PTSD-Checklist 5 | Visit 1 (Week 1/screening), Visit 2 (Week 2/Randomization/Baseline), Visit 3 (Week 3), Visit 4 (Week 4), Visit 5 (Week 5), Visit 6 (Week 6)
  The PCL-5 is a 20-item self-report measure that assesses the 20 DSM-5 symptoms of PTSD. A total symptom severity score (range - 0-80) can be obtained by summing the scores for each of the 20 items. Scores of 31-33 or higher suggests potential benefit from PTSD treatment. Scores lower than 31-33 may indicate the patient either has subthreshold symptoms of PTSD or does not meet criteria for PTSD.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer C Naylor, PhD, Principal Investigator — Durham VA Medical Center, Durham, NC; Christine E. Marx, MD MA, Principal Investigator — Durham VA Medical Center, Durham, NC
Locations (1):
- Durham VA Medical Center, Durham, NC, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No